CLINICAL TRIAL: NCT05147467
Title: A Single-arm, Pivotal Registration Phase II Study of the Efficacy and Safety of APG-2575 Monotherapy in Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: Study of APG-2575 in Patients With Relapsed/Refractory CLL/SLL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG2575CC201
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; APG-2575
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lisaftoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APG-2575 single agent in Relapse/Refractory CLL/SLL (Experimental): APG-2575 orally once daily at 600mg dose levels, every 28 days as a cycle.
  Interventions: Drug: APG2575

INTERVENTIONS:
Drug: APG2575 — APG-2575 orally once daily at 600mg dose levels, every 28 days as a cycle.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of APG-2575 single agent in patients with relapsed/refractory CLL/SLL.

DETAILED DESCRIPTION:
This is an single-arm, open-label, multi-center, pivotal registration Phase II study of efficacy and safety of APG-2575 as a single agent in relapsed/refractory CLL/SLL patients.

This study plans to enroll approximately 75 CLL/SLL subjects who have failed or are intolerant to prior immunochemotherapy and BTK inhibitor therapy. Eligible subjects will receive APG-2575 600mg, orally administered once daily (QD), within half an hour of a low-fat meal, for a cycle of 28 days. Participants will continue to accept APG - 2575 until the "end of treatment" that are consistent with the provisions in the solution of the termination of any specified standards.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet each of the following inclusion criteria are eligible to participate in this study:

1. Age ≥18 years old.
2. Pathologically confirmed CLL/SLL according to the 2018 revised IWCLL NCI-WG guidelines, subject with measurable lesions or splenomegaly due to CLL.
3. Expected survival is at least 12 weeks.
4. Refractory, recurrent, or intolerant to BTK inhibitors and immunochemotherapy,or first-line treatment with BTK inhibitors fails and is not suitable for immunochemotherapy.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): 0 -2.
6. Ability to understand and willingness to sign a written informed consent form approved by EC committee (the consent form must be signed by the patient prior to any screening or study-specific procedures).
7. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

1. Prior history of allogeneic hematopoietic stem cell transplantation, adoptive cell immunotherapy or autologous hematopoietic stem cell transplantation within 24 months.
2. Failure to recover adequately, at the discretion of the investigator, from prior surgical procedures. Patients who have had major surgery within 28 days from study entry, and patients who have had minor surgery within 14 days of study entry.
3. Received Bcl-2 inhibitor treatment.
4. Invasive NHL transformation or central nervous system (CNS) involvement has occurred.
5. Pregnancy or lactation, or pregnancy is expected during the study period or within 3 months after the last administration of treatment.
6. Within 2 years before entering the study, the subject had a history of active malignant tumors other than CLL / SLL, except that:

   * Fully treated cervical carcinoma in situ;
   * Completely resected basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
   * Confinement and resection of previously cured malignancies (or other treatment).
7. Any other condition or circumstance that would, at the discretion of the investigator, make the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 9 months after the last subject enrolled.
  ORR is defined by Complete Remission (CR)+ CR with incomplete marrow recovery (CRi) + Partial Remission (PR) (according to NCI-WG CLL(2018)) and by CR+PR ( according to Lugano (2014)).Response will be evaluated every 2 cycles (8 weeks) till complete treatment or one month after last dose.

SECONDARY OUTCOMES:
Progress Free Survival (PFS) | Up to 9 months after the last subject enrolled.
  PFS is defined as the time from the first administration to disease progression(PD) or death from any cause.
Time To Progression (TTP) | Up to 9 months after the last subject enrolled.
  TTP is defined as the time from the first administration to PD.
Time To Response (TTR) | Up to 9 months after the last subject enrolled.
  TTR is defined as the time from the first administration to the subjects' first CR, CRi, or PR.
Duration of Response (DOR) | Up to 9 months after the last subject enrolled.
  DOR is defined as the time from the subject's first CR, CRi, or PR to PD or death from any cause.
Overall Survival (OS) | Up to 9 months after the last subject enrolled.
  OS is defined as the time from the first administration to death.
the time of half absolute lymphocyte value (ALC) | Up to 9 months after the last subject enrolled.
  The time of half absolute lymphocyte value (ALC) is defined as the time from the first administration to 50% reduction of ALC of baseline.
Adverse events | Up to 9 months after the last subject enrolled.
  Adverse events (AE) and serious adverse events (SAE) will be graded according to NCI CTCAE Version 5.0.
Maximum plasma concentration (Cmax) | Up to 4 cycles (each cycle is 28 days).
  Maximum plasma concentration (Cmax) will be assessed on all participants with APG-2575 treatments.
Area under the plasma concentration versus time curve (AUC) | Up to 4 cycles (each cycle is 28 days).
  Area under the plasma concentration versus time curve (AUC) will be assessed on all participants with APG-2575 treatments.

OTHER OUTCOMES:
Minimal Residual Disease (MRD) negative rate | Up to 9 months after the last subject enrolled.
  To observe the proportion of subjects with MRD negative status in bone marrow, peripheral blood, one or both.
Bcl-2 expression | Up to 9 months after the last subject enrolled
  Potential biomarkers to be evaluated included the association of Bcl-2 expression with the efficacy of APG-2575 monotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Director — Ascentage Pharma Group Inc.; Jianyong Li, M.D., Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (11):
- China (11):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affilated Hospital of Soochow University, Suzhou, Jiangsu
  - People's hospital of Jiangsu Province, Suzhou, Jiangsu
  - The First Affilated Hospital of Nanchang University, Nanchang, Jiangxi
  - Institute of blood transfusion of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou, Zhejiang